CLINICAL TRIAL: NCT04980014
Title: Post-Marketing Surveillance Study on NesinaAct Tablet® Use Among Type 2 Diabetes Mellitus Patients in Korea
Brief Title: A Post-Marketing Surveillance Study on NesinaAct® Tablet Use Among Type 2 Diabetes Mellitus Participants in Korea
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Alogliptin-Pio-5002
Record Dates: First submitted 2021-07-26; First posted 2021-07-28 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NesinaAct® Tablet: Participants with a diagnosis of Type 2 Diabetes who took NesinaAct® tablet, a fixed dose combination of alogliptin along with pioglitazone, as prescribed by the physician, are observed in this study.
  Interventions: Drug: NesinaAct® Tablet

INTERVENTIONS:
Drug: NesinaAct® Tablet — NesinaAct® tablet is a fixed dose combination (FDC) of alogliptin benzoate with pioglitazone HCl.

SUMMARY:
The purpose of this post marketing surveillance (PMS) study is to estimate the proportion of all adverse events (AEs) including serious adverse events (SAEs) and serious adverse drug reactions (SADRs) in participants who are treated for type 2 diabetes mellitus under NesinaAct® tablet therapy (alogliptin/pioglitazone) once daily by physicians in the real-world clinical practice setting over a period of 26 weeks.

DETAILED DESCRIPTION:
The drug being tested in this survey is called NesinaAct® tablet. A surveillance is planned to examine safety and effectiveness of NesinaAct® tablet therapy in participants who are being treated for type 2 diabetes mellitus.

The study will enroll approximately 730 patients.

The study observes percentage of participants with adverse events (AEs) including serious adverse events (SAEs) and serious adverse drug reactions (SADRs) administered a dose of NesinaAct® tablet (alogliptin/pioglitazone) once daily as prescribed by the physician in routine practice over a period of 26 weeks.

This multi-center trial is conducted in a total of 19 sites in Korea.

The data is collected between October 2 2015 to August 30 2019 from the re-examination period up to 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants inadequately controlled on diet and exercise.
* Participants inadequately controlled on metformin alone.
* Participants inadequately controlled on pioglitazone alone.
* Participants inadequately controlled on metformin and pioglitazone combination therapy.
* Participants switching from alogliptin co-administered with pioglitazone.

Exclusion Criteria:

* Participants treated with study drug outside of the locally approved label in Korea.
* Participants with contraindication for the use of study drug (as described in the Korean product label).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with type 2 diabetes mellitus (T2DM) will be observed.
Sampling Method: Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- South Korea (8):
  - Busan
  - Chuncheon
  - Daejeon
  - Gangneung-si
  - Goyang-si
  - Jeonju
  - Seongam
  - Seoul

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this Post-Marketing Surveillance study at 19 investigative sites in Korea from 2 October 2015 to 30 August 2019 from the re-examination period.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes who took NesinaAct® Tablet, as prescribed by the physician, were enrolled in this study.
Groups:
- NesinaAct® Tablet: Participants with a diagnosis of Type 2 Diabetes who took NesinaAct® tablet, a fixed dose combination of alogliptin along with pioglitazone, as prescribed by the physician, were observed in this study.
Period: Overall Study
Arm/Group | NesinaAct® Tablet
Started | 730
Safety Analysis Set | 655
Effectiveness Analysis Set | 482
Completed | 655
Not Completed | 75
Not completed — Participants who are Duplicated | 1
Not completed — Follow-up Failure | 13
Not completed — Participants who did not Receive NesinaAct® Tablet | 2
Not completed — Participants who Have Been Administered NesinaAct® Tablet prior to the consent | 2
Not completed — Participants who Violated Inclusion/Exclusion Criteria | 57

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who were treated with NesinaAct® tablet at least once and completed the follow-up for safety.
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 655
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.32 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 400
  Male | 255
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 655
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Korea, Republic Of | 655

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) and Serious Adverse Drug Reactions (SADRs)
Description: An SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Serious ADRs are defined as SAEs that are, in the investigator's opinion, of causal relationship to the study treatment. 95% Confidence Interval was calculated using exact method.
Time Frame: First dose of surveillance drug treatment to within 30 days after the end of the treatment (up to 153 weeks)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 655
percentage of participants
  SAEs | 0.15 [0.00 to 0.85]
  SADRs | 0.00 [0.00 to 0.56]

2. Primary Outcome: Percentage of Participants With Unexpected Adverse Events (AEs) and Adverse Drug Reactions (ADRs) Not Mentioned in Precautions
Description: An AE is any and all undesirable or unintended signs (including abnormal clinical laboratory values), symptoms, or disease that are incurred when the drug is administered, and is not related to causal relationship with the drug. An ADR is a harmful and unintended reaction resulting from usual administration and use of the drug, whose causal relationship with the drug cannot be excluded, and if causal relationship with the drug is unknown among AEs reported spontaneously, it is regarded as ADR. An unexpected ADR is an ADR with difference in the nature or severity, specificity, or the outcome, compared to the product licensure/notification of the drug. 95% Confidence Interval was calculated using exact method.
Time Frame: First dose of surveillance drug treatment to within 30 days after the end of the treatment (up to 153 weeks)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 655
percentage of participants
  Unexpected AEs | 4.58 [3.11 to 6.47]
  Unexpected ADRs | 1.22 [0.53 to 2.39]

3. Primary Outcome: Percentage of Participants With Expected/Already Known ADRs at Week 13
Description: An ADR is a harmful and unintended reaction resulting from usual administration and use of the drug, whose causal relationship with the drug cannot be excluded, and if causal relationship with the drug is unknown among AEs reported spontaneously, it is regarded as ADR. Expected/already known ADRs are those listed in product licensure/notification of the drug. Data is reported as per duration of study drug treatment for this outcome measure from administration start date to AE onset date. 95% Confidence Interval was calculated using exact method.
Time Frame: Week 13
Population: Safety Analysis Set included participants who were treated with NesinaAct® tablet at least once and completed the follow-up for safety, with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 653
percentage of participants | 1.99 [1.06 to 3.38]

4. Primary Outcome: Percentage of Participants With Expected/Already Known ADRs at Week 26
Description: as for outcome 3
Time Frame: Week 26
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 515
percentage of participants | 0.19 [0.00 to 1.08]

5. Primary Outcome: Percentage of Participants With Expected/Already Known ADRs at Week 39
Description: as for outcome 3
Time Frame: Week 39
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 341
percentage of participants | 0.00 [0.00 to 1.08]

6. Primary Outcome: Percentage of Participants With Expected/Already Known ADRs at Week 52
Description: as for outcome 3
Time Frame: Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 108
percentage of participants | 0.93 [0.02 to 5.05]

7. Primary Outcome: Percentage of Participants With Expected/Already Known ADRs at Week 153
Description: as for outcome 3
Time Frame: Week 153
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 10
percentage of participants | 0.00 [0.00 to 30.85]

8. Primary Outcome: Percentage of Participants With Non-serious ADRs
Description: An ADR is a harmful and unintended reaction resulting from usual administration and use of the drug, whose causal relationship with the drug cannot be excluded, and if causal relationship with the drug is unknown among AEs reported spontaneously, it is regarded as ADR. 95% Confidence Interval was calculated using exact method.
Time Frame: First dose of surveillance drug treatment to within 30 days after the end of the treatment (up to 153 weeks)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 655
percentage of participants | 3.36 [2.12 to 5.04]

9. Primary Outcome: Percentage of Participants With Abnormal Laboratory Findings Reported as AEs
Description: Presence and absence of significant data in laboratory results were recorded. 95% Confidence Interval was calculated using exact method.
Time Frame: First dose of surveillance drug treatment to within 30 days after the end of the treatment (up to 153 weeks)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 655
percentage of participants
  Hyperglycaemia | 0.46 [0.09 to 1.33]
  Weight Increase | 0.31 [0.04 to 1.10]
  Diabetes Mellitus Aggravated | 0.15 [0.00 to 0.85]
  Hyperlipaemia | 0.15 [0.00 to 0.85]
  Sugar Blood Level Increase | 0.15 [0.00 to 0.85]
  Vitamin D Deficiency | 0.15 [0.00 to 0.85]

10. Secondary Outcome: Change From Baseline in Haemoglobin A1c (HbA1c) Levels
Description: HbA1c are glycated haemoglobin or amount of glucose attached to haemoglobin.
Time Frame: Baseline, Weeks 13 and 26
Population: Participants from the Effectiveness Analysis Set, included participants who completed NesinaAct® tablet treatment for more than 13 weeks and performed Final effectiveness assessment according to the investigator's clinical discretion, with data available for analyses. Number analyzed are participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 465
percentage of HbA1c
  Baseline | 7.90 (1.49)
  Change from Baseline at Week 13: number analyzed (Participants) | 347
  Change from Baseline at Week 13 | -0.93 (1.36)
  Change from Baseline at Week 26: number analyzed (Participants) | 201
  Change from Baseline at Week 26 | -1.40 (1.62)

11. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Time Frame: Baseline, Weeks 13 and 26
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 440
g/dL
  Baseline | 170.75 (46.65)
  Change from Baseline at Week 13: number analyzed (Participants) | 317
  Change from Baseline at Week 13 | -25.26 (40.44)
  Change from Baseline at Week 26: number analyzed (Participants) | 177
  Change from Baseline at Week 26 | -33.49 (43.18)

12. Secondary Outcome: Change From Baseline in Total Cholesterol
Description: Total cholesterol is a measure of the total amount of cholesterol in the blood. It includes both low-density lipoprotein (LDL) cholesterol and high-density lipoprotein (HDL) cholesterol.
Time Frame: Baseline, Weeks 13 and 26
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 401
mg/dL
  Baseline | 182.51 (39.37)
  Change from Baseline at Week 13: number analyzed (Participants) | 293
  Change from Baseline at Week 13 | -13.14 (30.86)
  Change from Baseline at Week 26: number analyzed (Participants) | 162
  Change from Baseline at Week 26 | -8.64 (35.84)

13. Secondary Outcome: Change From Baseline in Low Density Lipoprotein-Cholesterol (LDL-C)
Time Frame: Baseline, Weeks 13 and 26
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 375
mg/dL
  Baseline | 104.65 (33.17)
  Change from Baseline at Week 13: number analyzed (Participants) | 275
  Change from Baseline at Week 13 | -7.85 (23.40)
  Change from Baseline at Week 26: number analyzed (Participants) | 153
  Change from Baseline at Week 26 | -8.28 (27.99)

14. Secondary Outcome: Change From Baseline in High Density Lipoprotein-Cholesterol (HDL-C)
Time Frame: Baseline, Weeks 13 and 26
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 385
mg/dL
  Baseline | 47.18 (10.46)
  Change from Baseline at Week 13: number analyzed (Participants) | 280
  Change from Baseline at Week 13 | 2.36 (6.61)
  Change from Baseline at Week 126: number analyzed (Participants) | 151
  Change from Baseline at Week 126 | 1.90 (7.02)

15. Secondary Outcome: Change From Baseline in Body Weight
Time Frame: Baseline, Weeks 13 and 26
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 530
kg
  Baseline | 69.98 (11.73)
  Change from Baseline at Week 13: number analyzed (Participants) | 223
  Change from Baseline at Week 13 | -0.67 (2.01)
  Change from Baseline at Week 26: number analyzed (Participants) | 110
  Change from Baseline at Week 26 | -0.48 (2.60)

16. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Time Frame: Baseline, Weeks 13 and 26
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 547
mm Hg
  Baseline | 128.20 (12.52)
  Change from Baseline at Week 13: number analyzed (Participants) | 360
  Change from Baseline at Week 13 | -0.88 (11.48)
  Change from Baseline at Week 26: number analyzed (Participants) | 226
  Change from Baseline at Week 26 | -1.66 (12.44)

17. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Time Frame: Baseline, Weeks 13 and 26
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | NesinaAct® Tablet
Number analyzed (Participants) | 547
mm Hg
  Baseline | 79.84 (10.98)
  Change from Baseline at Week 13: number analyzed (Participants) | 360
  Change from Baseline at Week 13 | -1.40 (9.75)
  Change from Baseline at Week 26: number analyzed (Participants) | 226
  Change from Baseline at Week 26 | -0.34 (9.32)

ADVERSE EVENTS:
Time Frame: First dose of surveillance drug treatment to within 30 days after the end of the treatment (up to 153 weeks)
Description: Safety Analysis set included participants who were treated with NesinaAct® tablet at least once and completed the follow-up for safety.
Arm/Group | NesinaAct® Tablet
All-Cause Mortality (participants affected / at risk) | 0/655
Serious Adverse Events (participants affected / at risk) | 1/655
Other Adverse Events (participants affected / at risk) | 0/655
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NesinaAct® Tablet (N=655)
Tendon Rupture (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT04980014/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT04980014/SAP_001.pdf